CLINICAL TRIAL: NCT06006169
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of BL-B01D1 Monotherapy, SI-B003 Monotherapy and BL-B01D1+SI-B003 Combination Therapy (BL-B01D1+SI-B003) in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma and Other Solid Tumors
Brief Title: A Study of BL-B01D1, SI-B003 and BL-B01D1+SI-B003 in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma and Other Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-SI-B003-201-03
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-B01D1, SI-B003 or BL-B01D1 + SI-B003 therapy in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-B01D1; Drug: SI-B003

INTERVENTIONS:
Drug: BL-B01D1 — BL-B01D1 was administered by intravenous infusion on D1, D8, or D1 in 3-week cycles.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: SI-B003 — SI-B003 was administered intravenously every 3 weeks (Q3W).

SUMMARY:
This phase II study is designed to investigate the efficacy and safety of BL-B01D1 monotherapy, SI-B003 monotherapy, and BL-B01D1+SI-B003 combination therapy in patients with recurrent or metastatic head and neck squamous cell carcinoma and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects voluntarily participated in the study and signed informed consent.
2. Male or female aged ≥18 years and ≤75 years.
3. Expected survival time ≥3 months.
4. ECOG 0-1.
5. Patients with recurrent or metastatic head and neck squamous cell carcinoma (non-nasopharyngeal carcinoma) confirmed by histopathology and/or cytology:

   1. Cohort_A, B, and Cohort_C Stage I patients who had failed or were intolerant to 1 or more lines of systemic therapy for recurrent or metastatic HNSCC (non-nasopharyngeal carcinoma);
   2. Cohort_C Stage II patients who had not received any previous systemic antitumor therapy (other than induction chemotherapy, neoadjuvant, or adjuvant therapy) for recurrent or metastatic HNSCC (non-nasopharyngeal); Treatment failure was defined as disease progression during or after systemic antitumor therapy.

   Intolerance refers to the refusal of patients to continue the original regimen due to grade 3-4 adverse reactions after receiving standard treatment.

   Note: Recurrence or disease progression within 6 months after the last chemotherapy of multimodal therapy was considered as the first line of treatment.
6. Consent to provide archival tumor tissue specimens (10-12 unstained sections (anti-slip) surgical specimens (thickness 4-5μm)) or fresh tissue samples from primary or metastatic lesions within 3 years. If participants cannot provide tumor tissue samples, they can be enrolled if they meet other inclusion and exclusion criteria after the evaluation of the investigator.
7. Must have at least one measurable lesion according to RECIST v1.1 definition; Lesions that had been previously treated with radiation could be included in a measurable lesion only if there was definite disease progression after radiation therapy.
8. No blood transfusions and no use of cell growth factors and/or platelet-raising drugs during the 14 days prior to the screening period must be allowed, and the organ function level must meet the following criteria:

   1. Blood routine: hemoglobin (HGB) ≥ 90g/L; Absolute neutrophil count (NEUT) ≥ 1.5×10 9 /L; Platelet count (PLT) ≥ 100×10 9 /L;
   2. Renal function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula).
   3. Liver function: total bilirubin (TBIL≤1.5 ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were all ≤2.5 ULN, and AST and ALT were both ≤5.0 ULN when liver metastasis was present;
   4. coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5ULN;
   5. no severe cardiac dysfunction with left ventricular ejection fraction ≥50%;
   6. proteinuria ≤2+ or ≤1000mg/24h.
9. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic laboratory abnormalities such as ALP elevation, hyperuricemia, and hyperglycemia, as judged by the investigator, and toxicity without safety risk, such as alopecia, grade 2 peripheral neurotoxicity, or decreased hemoglobin ≥90g/L, as judged by the investigator).
10. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the start of treatment, the serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the whole treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Prior treatment with an ADC drug with a topoisomerase I inhibitor as a toxin.
2. Antineoplastic therapy, including chemotherapy, biologic therapy, immunotherapy, definitive radiotherapy, major surgery (investigator-defined), or targeted therapy (including small-molecule tyrosine kinase inhibitors), has been administered within 4 weeks or 5 half-life cycles (whichever is shorter) before the first dose; Oral fluorouracil drugs such as S-1, capecitabine, or palliative radiotherapy within 2 weeks before the first dose.
3. Non-squamous cell tissue confirmed by histopathology and/or cytology must be excluded.
4. Cohort_C Stage II patients who had received any previous systemic therapy for recurrent or metastatic HNSCC (other than induction chemotherapy, adjuvant or neoadjuvant therapy) were excluded.
5. Cohort_C with a history of immunotherapy and grade ≥3 irAE or grade ≥2 immune-related myocarditis, excluded.
6. Cohort_C cohort_c who had received immunomodulatory drugs (including but not limited to thymosin, interleukin-2, interferon, etc.) within 14 days before the first dose of study drug was excluded.
7. Systemic corticosteroids (> 10mg/ day of prednisone, or the equivalent of another corticosteroid) are required within 2 weeks before the first dose of the study dose; Exceptions were inhaled or topical corticosteroids or physiological replacement doses of corticosteroids for adrenal insufficiency.
8. A history of immunotherapy with grade ≥3 irAE or grade ≥2 immune-related myocarditis must be excluded.
9. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

   1. severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias or Ⅲ degree atrioventricular block requiring clinical intervention;
   2. prolonged QT interval at rest (QTc > 450 msec in men or QTc > 470 msec in women);
   3. myocardial infarction, unstable angina, cardiac angioplasty or stent implantation, coronary artery/peripheral artery bypass grafting, New York Heart Association (NYHA) class III or IV congestive heart failure, cerebrovascular accident, or transient ischemic attack within 6 months before the first dose.
10. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory intestinal diseases and Hashimoto's thyroiditis, etc., excluding type I diabetes mellitus, hypothyroidism that can be controlled only by replacement therapy, and skin diseases without systemic treatment (such as vitiligo and psoriasis).
11. Other malignant tumors that have progressed or require treatment within 3 years before the first dose, except for radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, radical resection of carcinoma in situ, such as carcinoma in situ of the breast, prostate cancer; Notes: Patients with localized low-risk prostate cancer (defined as stage ≤T2a, Gleason score ≤6, and PSA < 10ng/mL at prostate cancer diagnosis (as measured) who had received radical treatment and no biochemical recurrence of prostate specific antigen (PSA) were eligible to participate in this study).
12. A history of (non-infectious) interstitial lung disease (ILD)/pulmonary inflammation requiring steroid treatment, or current ILD/ pulmonary inflammation, or suspected ILD/ pulmonary inflammation that cannot be ruled out by imaging at screening.
13. Before starting the study treatment, there are:

    1. Poorly controlled diabetes (fasting blood glucose ≥ 13.3 mmol/L)
    2. Poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
    3. History of hypertensive crisis or hypertensive encephalopathy.
14. Unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening; Infusion-related thrombosis was excluded.
15. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases). Patients who had received treatment for brain metastases (radiotherapy or surgery; Patients with stable brain metastases who had stopped radiotherapy or surgery 28 days before the first dose were eligible. Patients with cancerous meningitis (meningeal metastases) were excluded even if they were treated and judged to be stable. Stable disease was defined as being asymptomatic, in stable condition, and not requiring steroid therapy for more than 4 weeks before starting study treatment.
16. Patients with pleural effusion, pericardial effusion or ascites with clinical symptoms or requiring repeated drainage.
17. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any excipients of BL-B01D1.
18. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT).
19. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > 103 IU/ml) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > detection limit).
20. Active infections requiring systemic therapy, such as severe pneumonia, bacteremia, sepsis, etc.
21. Had participated in another clinical trial within 4 weeks before the first dose (calculated from the time of the last dose).
22. Persons with a history of psychotropic drug abuse and inability to quit or mental disorders.
23. Other circumstances considered by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, Principal Investigator — Fudan University; Dongmei Ji, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China